CLINICAL TRIAL: NCT02326168
Title: A Study Evaluating the Safety and Tolerability of Percutaneous Vaccination Prior to Intravesical Instillation of Bacillus Calmette-Guerin (BCG) Mycobacteria for Non-Muscle Invasive Bladder Cancer
Brief Title: PRIME: Pilot Study Evaluating Percutaneous Vaccination of BCG for Bladder Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Robert Svatek, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140005
Record Dates: First submitted 2014-12-05; First posted 2014-12-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non-muscle invasive bladder cancer (Experimental): Every patient meeting eligibility criteria will receive a standard WHO adult potency Bacillus Calmette-Guerin (BCG) immunization (1cc/50mg live mycobacilli) in the right or left deltoid. Following a 19 - 31day wait period after BCG vaccination patients will then receive standard strength BCG intravesical therapy returning once a week for 6 consecutive weeks. Cystoscopy will be performed at 3 and 6 months.
  Interventions: BCG immunization in deltoid and BCG intravesical therapy once a week for 6 weeks.
  Interventions: Drug: Bacillus Calmette-Guerin (BCG)

INTERVENTIONS:
Drug: Bacillus Calmette-Guerin (BCG) — Intravesical instillation for non-muscle invasive bladder cancer
  Other Names: Tice BCG

SUMMARY:
Approximately 25 subjects will be enrolled and receive a standard WHO adult potency BCG immunization (1cc/50mg live mycobacilli) in the deltoid. Following a wait period after BCG vaccination, patients will then receive standard strength BCG intravesical therapy once a week for a total of 6 weeks. The BCG is instilled and held in the bladder for approximately 2 hours. While the BCG is retained in the bladder the patient should be repositioned every 30 minutes to maximize bladder surface exposure to the agent. Patients will undergo a cystoscopy every 3 months following most recent TURBT. Study duration last approximately 6 months.

DETAILED DESCRIPTION:
Approximately 25 subjects will receive a standard WHO adult potency BCG immunization (1cc/50mg live mycobacilli) in the deltoid. Following a wait period after BCG vaccination, patients will then receive standard strength BCG intravesical therapy once a week for a total of 6 weeks. The BCG is instilled and held in the bladder for approximately 2 hours. While the BCG is retained in the bladder the patient should be repositioned every 30 minutes to maximize bladder surface exposure to the agent. Patients will undergo a cystoscopy every 3 months following most recent TURBT. Study duration last approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

The patient must:

* Be 18 years of age or older
* Be able to give informed consent
* Have newly diagnosed or recurrent multi-focal Ta, Large Ta, High Grade Ta, CIS or T1 Bladder Cancer
* Determined by treating urologist to be a good candidate for BCG Induction Therapy
* Have an adequate marrow function (defined as white blood cells greater than 1.5 x 103/µl (or 1,500 cells/mm3) and platelets greater than 150,000 cells/mm3; these results can be within last 60 days from the day of signing informed consent

Exclusion Criteria:

The patient cannot:

* Be less than18 years of age
* Unable to give informed consent
* Have a history of muscle invasive bladder cancer
* Be self-reported to be immune-compromised (HIV, chronic immunomodulators, chronic corticosteroids)
* Have a history of tuberculosis and/or received BCG Percutaneous Vaccination
* Pregnant or planning to become pregnant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
BCG response | 3 months after baseline
  Percentage of patients with complete response at 3 months following therapy of combined percutaneous vaccination with TICE percutaneous Bacillus Calmette-Guerin (BCG) vaccine combined with standard protocol intravesical induction BCG vaccine for patients with non-muscle invasive transitional cell carcinoma of the bladder.

SECONDARY OUTCOMES:
PPD conversion | 3 months from BCG vaccination
  PPD conversion from negative to positive (defined as ≥ 10 mm induration at 48-72 hours following PPD placement).

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Svatek, MD, Principal Investigator — Unv Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center, San Antonio, Texas, United States